CLINICAL TRIAL: NCT01934738
Title: A Phase 1, Double Blind (3rd Party Open) Randomized, Placebo Controlled, Dose Escalation Study to Investigate the Safety, Tolerability and Pharmacokinetics of Repeat Doses of PF-06273340 in Healthy Subjects
Brief Title: A Study to Evaluate Safety, Toleration and Time Course of Plasma Concentration of Multiple Oral Doses of PF-06273340 in Healthy Subjects of Two AgeGroups, Aged 18-55 Years (Group 1) and Aged 56-75 Years (Group 2)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: B5261002
Record Dates: First submitted 2013-08-30; First posted 2013-09-04 (Estimated); Last update posted 2014-03-11 (Estimated); Status verified 2014-03

CONDITIONS: Healthy
Keywords: Multiple dose; safety; tolerability; PK
MeSH Terms: interventions — PF-06273340

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- Group 1: Cohort 1 (Experimental)
  Interventions: Drug: PF-06273340; Drug: Placebo
- Group 1: Cohort 2 (Experimental)
  Interventions: Drug: PF-06273340; Drug: Placebo
- Group 1: Cohort 3 (Experimental)
  Interventions: Drug: PF-06273340; Drug: Placebo
- Group 2: Cohort 4 (Experimental)
  Interventions: Drug: PF-06273340; Drug: Placebo
- Group 1: Cohort 5 (Experimental)
  Interventions: Drug: PF-06273340; Drug: Placebo
- Group 2: Cohort 6 (Experimental)
  Interventions: Drug: PF-06273340; Drug: Placebo

INTERVENTIONS:
Drug: PF-06273340 — Tablets, 100 mg TID, 14 days
  Arms: Group 1: Cohort 1
Drug: Placebo — Tablets, TID, 14 days
  Arms: Group 1: Cohort 1
Drug: PF-06273340 — Tablets, to be decided dose, TID or titration, 14 days
  Arms: Group 1: Cohort 2
Drug: Placebo — Tablets, TID or titration, 14 days
  Arms: Group 1: Cohort 2
Drug: PF-06273340 — Tablets, to be decided dose, TID or titration, 14 days
  Arms: Group 1: Cohort 3
Drug: Placebo — Tablets, TID or titration, 14 days
  Arms: Group 1: Cohort 3
Drug: PF-06273340 — Tablets, to be decided dose, TID or titration, 14 days
  Arms: Group 2: Cohort 4
Drug: Placebo — Tablets, TID or titration, 14 days
  Arms: Group 2: Cohort 4
Drug: PF-06273340 — Tablets, to be decided dose, TID or titration, 14 days
  Arms: Group 1: Cohort 5
Drug: Placebo — Tablets, TID or titration, 14 days
  Arms: Group 1: Cohort 5
Drug: PF-06273340 — Tablets, to be decided dose, TID or titration, 14 days
  Arms: Group 2: Cohort 6
Drug: Placebo — Tablets, TID or titration, 14 days
  Arms: Group 2: Cohort 6

SUMMARY:
The purpose of this study is to investigate safety, toleration and time course of plasma concentration of multiple oral doses of PF-06273340 for 14 days in healthy subjects of two age groups, aged 18-55 years (Group 1) and aged 56-75 years (Group 2)

ELIGIBILITY:
Inclusion Criteria:

* For Group 1 specific: Healthy male and/or female subjects of non-childbearing potential between the ages of 18 and 55 years, inclusive (Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and pulse rate measurement, 12-lead ECG and clinical laboratory tests).
* For Group 2 specific: Healthy male and/or female subjects of non-childbearing potential between the ages of 56 and 75 years, inclusive. Subjects must be in reasonably good health as determined by the investigator based on a detailed medical history, full physical examination (including blood pressure and pulse rate measurement), 12-lead ECG and clinical laboratory tests. Subjects with mild, chronic, stable disease (eg, osteoarthritis) may be enrolled if deemed medically prudent by the investigator. In order to ensure an age range relevant to the osteoarthritis (OA) population, at least 50% of the subjects enrolled in these cohorts must be 60 years of age and above at Screening.
* For Group 2 specific: Subjects taking daily prescription or non-prescription medications for management of acceptable chronic medical conditions must be on a stable dose of these, as defined by non change in dose for the 3 months prior to the first dose of study medication and no planned changes during the conduct of the study.

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).
* Any condition possibly affecting drug absorption (eg, gastrectomy).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2013-10; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) | 14 days
Area Under the Curve from Time Zero to end of dosing interval (AUCtau) | 14 days
Time to Reach Maximum Observed Plasma Concentration (Tmax) | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Brussels, Belgium

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B5261002&StudyName=A%20Study%20to%20Evaluate%20Safety%2C%20Toleration%20and%20Time%20Course%20of%20Plasma%20Concentration%20of%20Multiple%20Oral%20Doses%20of%20PF-06273340%20in%20Healthy%20Subj